CLINICAL TRIAL: NCT03182712
Title: Effects of n-3 Fatty Acids and Vitamin E Supplementation Upon Oxidative Stress, Inflammation and Metabolic Parameters in Type 2 Diabetic Subjects at Rest and After an Acute High Intensity Exercise Bout
Brief Title: n-3 Fatty Acid Effects in T2DM After Acute High Intensity Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Maurício Krause, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HCPA 06-222
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The selected subjects were referred to the University laboratory. During their first visit, the subjects were submitted to perform the first high intensity sub-maximal test. In the same day, volunteers received the supplementation capsules that should be taken throughout eight weeks, as described in the supplementation section.
  The subjects were randomly assigned to two groups: (1) group placebo and (2) n-3 PUFA group. After the supplementation period, all subjects reported back to hospital to biochemical testing and thereafter to the university exercise laboratory for the second high intensity sub-maximal test, following the same protocol described above.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- n-3 PUFA Group (Experimental): Subjects receiving n-3 PUFA (capsules containing 180 mg of eicosapentaenoic acid, 120 mg of docosahexaenoic acid and 2 mg of vitamin E). Three capsules were ingested daily for eight weeks.
  Interventions: Dietary Supplement: n-3 PUFA Group
- Placebo Group (Placebo Comparator): Subjects receiving gelatin capsules (500mg). Three capsules were ingested daily for eight weeks.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: n-3 PUFA Group — Participants received n-3 PUFA capsules (capsules containing 180 mg of eicosapentaenoic acid, 120 mg of docosahexaenoic acid and 2 mg of vitamin E). Three capsules were ingested daily for eight weeks, distributed between breakfast, lunch and dinner.
  Arms: n-3 PUFA Group
Dietary Supplement: Placebo Group — Participants received capsules containing 500 mg of gelatin.Three capsules were ingested daily for eight weeks, distributed between breakfast, lunch and dinner.
  Arms: Placebo Group

SUMMARY:
The aim of this study was to verify the effect of a combined supplementation [n-3 PUFA (known to induce anti-inflammatory effects) plus vitamin E (known for its antioxidant properties)] on lipidic, glycemic, redox status and inflammatory parameters in type 2 diabetic patients. In addition, considering that exercise, at high intensities, can induce a transient inflammatory state and increase oxidative stress (OS) markers, the investigators tested if our nutritional intervention could attenuate this response within this population (thus, using high intensity exercise as inductor of acute inflammatory/OS state).

DETAILED DESCRIPTION:
Herein the investigators tested the effect of eight weeks of omega-3 polyunsaturated fatty acid (n-3 PUFA) and vitamin E supplementation before and after an acute high intensity exercise bout on lipid profile, glycemic, redox and inflammatory parameters in type 2 diabetic (T2DM) patients. Thirty T2DM patients, without chronic complications, took part in this study. Blood and urine samples were collected after 12 h-fasting state for baseline biochemical analysis. Thereafter, subjects performed an incremental workload VO2max test on a cycle ergometer to determine the load of the high intensity submaximal exercise. On the following week, blood samples were collected before and immediately after the exercise test for measurements of oxidative stress (OS) and high-sensitivity C-reactive protein (hs-CRP). Afterwards, participants were randomly allocated into two groups: placebo (gelatin) and n-3 PUFA (capsules containing 180 mg of eicosapentaenoic acid, 120 mg of docosahexaenoic acid and 2 mg of vitamin E). Three capsules were ingested daily for eight weeks. Then, the examination protocol and the exercise test were repeated and the samples collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes
* Male and female
* Age between 40 and 60 years old.
* Must be able to do exercise

Exclusion Criteria:

* Smoking;
* Clinical diagnosis of kidney, pulmonary or heart diseases

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02-10 (Actual); Study Completion 2008-03-15 (Actual)

PRIMARY OUTCOMES:
Changes on hs-CRP (High-sensitivity C reactive protein) | Measured before the supplementation (baseline) and after eight weeks of supplementation
  Marker of inflammation expressed in mg/dL

SECONDARY OUTCOMES:
Changes on F2-isoprostanes | Measured before the supplementation (baseline) and after eight weeks of supplementation
  Marker of oxidative stress expressed in ng/mL
Changes on thiobarbituric acid reactivity | Measured before the supplementation (baseline) and after eight weeks of supplementation
  Marker of oxidative stress expressed in nmol/mL
Changes on Total Antioxidant activity | Measured before the supplementation (baseline) and after eight weeks of supplementation
  Marker of oxidative stress expressed in contains per minute

CONTACTS AND LOCATIONS:
Overall Officials: Rogério Friedman, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Clinical Hospital of Porto Alegre, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data, including body composition, inflammatory and oxidative stress markers and metabolites.

REFERENCES:
- [Derived] Fayh APT, Borges K, Cunha GS, Krause M, Rocha R, de Bittencourt PIH Jr, Moreira JCF, Friedman R, da Silva Rossato J, Fernandes JR, Reischak-Oliveira A. Effects of n-3 fatty acids and exercise on oxidative stress parameters in type 2 diabetic: a randomized clinical trial. J Int Soc Sports Nutr. 2018 Apr 23;15:18. doi: 10.1186/s12970-018-0222-2. eCollection 2018. PMID 29713249